CLINICAL TRIAL: NCT06859801
Title: A Multi-Center Observational Trial of Symptomatic, High-Risk Bone Metastases Treated with Percutaneous Ablation and Palliative Radiation Therapy
Acronym: TRIBUTE
Status: Not yet recruiting | Type: Observational
Sponsor: Society of Interventional Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: SIO-2025-01
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Bone Cancer Metastatic
MeSH Terms: interventions — Catheter Ablation; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Percutaneous Ablation — Percutaneous ablation is a minimally invasive alternative therapy for metastatic bone disease and can be used for destruction of nerves mediating pain signals, tumor destruction, decompression, or inhibition of tumor growth.
Radiation: Radiation Therapy — Radiation therapy (RT) is a widely accepted treatment for painful bone metastases and provides palliation of pain for patients.

SUMMARY:
The objective of this study is to evaluate real-world outcomes (e.g., pain, patient reported outcomes, skeletal related events, healthcare utilization, etc.) in patients treated with both percutaneous ablation and palliative radiation therapy (RT).

ELIGIBILITY:
Inclusion Criteria:

* 1. Skeletal metastasis with localized pain not controlled medically [recall within last 24 hours of worst pain ≥ 5 using the BPI]
* 2. Pain must be from one painful metastatic lesion involving the bone (additional less painful metastatic sites may be present). Extra-osseous extension of disease is allowed (must have some contact with the bone and be causing bone/tumor interface pain)
* 3. Lesions that are at high-risk of skeletal related events defined as follows:
* a. Minimum Spinal Instability Neoplastic Score (SINS) score ≥ 7 for lesions involving the spine
* b. Pelvic and appendicular lytic lesions with or without cortical breakthrough causing functional/mechanical pain
* 4. Target lesion amenable to percutaneous ablation with image guidance AND RT by specialists' review
* 5. No prior targeted radiation therapy or ablation to the index lesion
* 6. ECOG performance status 0-2
* 7. Age ≥ 21 years
* 8. Have signed the current approved informed consent form
* 9. Willing and able to answer follow-up Patient Reported Outcomes (PRO) surveys (e.g., PROMIS®, BPI, COST-FACIT, and OMED) for up to 12 months
* 10. Life expectancy > 3 months

Exclusion Criteria:

* 1. Any medical or personal condition that, in the opinion of the site investigator, may potentially compromise the safety or compliance of the patient, or may preclude the patient's successful completion of the clinical trial.
* 2. Target tumor involves a weight-bearing long bone of the lower extremity with the tumor causing > 50% loss of cortical bone [MIREL Score ≥ 7]
* 3. Skeletal lesions with unstable pathologic fractures requiring immediate surgical stabilization
* 4. Concurrent participation in other studies that could affect the primary endpoint
* 5. Target tumor causing clinical or imaging evidence of spinal cord compression

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with previously untreated symptomatic, high-risk skeletal metastases who are scheduled to be treated with percutaneous ablation combined with palliative RT as part of their normal Standard of Care (SOC).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain Response | 3 Months
  Combined partial and complete pain response rate using the Brief Pain Inventory (BPI), worst pain 24-hour recall, at 3 months following percutaneous ablation and palliative RT as defined by International Consensus on Palliative Radiotherapy Endpoints in clinical trials (ICPRE).
  • Partial response is defined as pain reduction of 2 or more at the treated site on a scale of 0 to 10 scale without analgesic increase, or analgesic reduction of 25% or more from Baseline without an increase in pain.
  • Complete response is defined as a pain score of 0 at the treated site with no concomitant increase in analgesic intake (stable or reducing analgesics in daily OMED).